CLINICAL TRIAL: NCT04943978
Title: Prospective Studies on the Immunopathogenesis of Fibrosis in Acute and Chronic Liver Diseases
Brief Title: Prospective Studies on Immunopathogenesis of Liver Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Edward Geissler, Head of Exp. Surgery, University of Regensburg
Other Study IDs: 13-257-101
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Chronic Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liver biopsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver disease: Patients with either acute or chronic liver disease

INTERVENTIONS:
Other:  — just observational blood and liver sampling
  Other Names: No Intervention

SUMMARY:
The immune system is thought to play a key role in the development of liver inflammation and subsequent liver fibrosis or cirrhosis.

In the case of viral hepatitis and autoimmune hepatitis, for example, numerous studies have focused on the acquired antigen-specific immunity. However, the liver is the site of increased occurrence of the components of the innate immune response (NK and NKT cells) and, in contrast to T cells, these T cells, these do not require antigen presentation.

Therefore, the present study was designed to determine which cellular components of the (NK, NKT, dendritic cells, macrophages) or the acquired immune response (CD4, CD8) or which network of immune cells is involved in the immunopathogenesis of progressive liver inflammation or the development of liver fibrosis.

The aim is to identify lymphocyte populations that exhibit either prognostically favorable or unfavorable characteristics. This should allow conclusions to be drawn for a more targeted and individualized therapy of the respective chronic liver diseases.

DETAILED DESCRIPTION:
In patients with acute liver inflammation (e.g., autoimmune hepatitis, viral hepatitis) or chronic inflammation (e.g., ethyltoxic, viral hepatitis, fatty liver, autoimmune hepatitis, colorectal liver metastases, HCC) or liver fibrosis, the cellular immune response will be prospectively investigated and compared with liver healthy control patients.

For this purpose, patients with known or unknown liver disease will be tested during inpatient stays or during a visit to the outpatient clinic after written consent has been obtained.

Blood is then processed for further immunological cell analyses and finally frozen in liquid nitrogen. If a liver biopsy is taken from the patient as part of the clinical diagnostics during an inpatient stay or if a liver biopsy or liver resection is performed during a procedure in the OR, tissue that is not required for diagnostic purposes should be frozen for further immunological cell analysis.

If patients undergoing elective surgery in the abdominal cavity are suspected of having a liver disease (e.g., altered liver parameters in the blood) and a wedge biopsy of the liver will be performed intraoperatively for diagnostics, tissue that is not required for diagnostic purposes should be prepared for further immunological cell analysis.

In addition, a part of the liver tissue obtained should be preserved for later genetic studies, e.g. in RNA-later.

In case of acute liver disease, further blood samples should be taken 48 and 96 h later and on weeks 1, 2, 4, 6, and 12, and after 6 and 12 months, respectively (or at the respective visits to the outpatient clinic).

For patients with chronic liver disease, blood should be re-collected during their regular visits at the outpatient clinic

In addition to patient history and medical information, the patients should also be regularly examined during the entire duration of the study and medical information, that are regularly collected during routine laboratory work ups (e.g. viral titers by quantitative PCR, liver enzymes and liver function) will be included.

To compare the immune responses, lymphocytes from patients without liver disease will be examined. will be investigated. Furthermore, healthy blood donors will be used as an additional control group.

ELIGIBILITY:
Inclusion Criteria:

Patients with chronic liver disease up to progressive cirrhosis (e.g. ethyltoxic, Viral hepatitis, fatty liver, autoimmune hepatitis, colorectal liver metastases, HCC).

Patients with elevated liver values undergoing elective abdominal surgery.

As comparison groups patients with acute hepatitis (e.g. viral or autoimmune genesis) and patients without liver disease.

Exclusion Criteria:

Age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic or acute liver disease undergoing surgery.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-02-01 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Liver fibrosis | Day 0
  Stage of liver fibrosis in histology (Ishak-score (1 - 6))
Liver Steatosis | Day 0
  Stage of liver steatosis in histology (NASH activity score (1 - 8))

SECONDARY OUTCOMES:
Survival | After 3 years
  Overall Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Surgery, University Hospital Regensburg, Regensburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Depending on data safety plan